CLINICAL TRIAL: NCT02302586
Title: Effects of Thoracic Paravertebral Blockade on Acute and Chronic Pain After Video Assisted Thoracoscopic Surgery (VATS) - A Randomized, Clinical Trial
Brief Title: Thoracic Paravertebral Blockade in Video Assisted Thoracoscopic Surgery (VATS)
Acronym: VATS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nuzhet Mert Senturk, MD, Prof, MD, Prof. Dr, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 46143867-1035
Record Dates: First submitted 2014-11-20; First posted 2014-11-27 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Pain, Postoperative
Keywords: Thoracic paravertebral block; Patient controlled analgesia; Video Assisted Thoracoscopic Surgery; Postoperative acute pain; Chronic pain
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — Bupivacaine; Analgesia, Patient-Controlled; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient Controlled Analgesia (IV PCA) (Active Comparator): Postoperative intravenous (IV) morphine PCA is being used for acute pain control: Basal infusion: 0.3 mg/kg/h Bolus: 1 mg, Lock-out time: 20 min, 4-h limit: 10-12,5 mg
  Interventions: Drug: Patient Controlled Analgesia (IV PCA)
- Thoracic Paravertebral Block (TPVB) (Active Comparator): Preoperative thoracic paravertebral block (TPVB) at 4 levels from T4 to T8 is being performed and total of 20 mL Bupivacaine 0.5% is deposited (5 mL per level by using landmark technique)
  Interventions: Drug: Thoracic paravertebral block (TPVB)

INTERVENTIONS:
Drug: Thoracic paravertebral block (TPVB) — Thoracic paravertebral block (TPVB) is being performed by injecting 5 mL of Bupivacaine 0.5% to 4 consecutive level of paravertebral spaces between T4 and T8 by using landmark technique
  Other Names: Bupivacaine
  Arms: Thoracic Paravertebral Block (TPVB)
Drug: Patient Controlled Analgesia (IV PCA) — IV morphine patient controlled analgesia (PCA) is being used in the postoperative period for 48 hours. Basal infusion: 0.3 mg/kg/h, Bolus: 1 mg, Lock-out time: 20 min, 4-h limit: 10-12,5 mg
  Other Names: Morphine
  Arms: Patient Controlled Analgesia (IV PCA)

SUMMARY:
Video-assisted thoracoscopic surgeries (VATS) include severe postoperative acute pain which is also a predictor of chronic pain. In this study, the investigators aim to compare the postoperative effects of thoracic paravertebral block (TPVB) and intravenous patient controlled analgesia (PCA) on the prevention of chronic pain of patients undergoing VATS.

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgeries (VATS) include significant postoperative acute and chronic pain because of trocar site tissue damages, intercostal nerve injuries and related inflammatory responses. Poorly controlled pain in the early postoperative period usually causes chronic pain, and also affects patients' physiotherapy, mobilization and daily function.

Our hypothesis in this study is 'thoracic paravertebral block (TPVB) is associated with an improvement in control of acute and chronic pain after VATS compared to systemic analgesia.

ELIGIBILITY:
Inclusion Criteria:

ASA I-III Patients who undergo Video-assisted thoracoscopic surgery (VATS) under GA

Exclusion Criteria:

Patients with difficult understanding the instructions for using PCA and/or pain scales Patients with contraindication to regional anesthesia Patients with significant neurologic, psychiatric or cognitive disorders History of substance abuse or chronic opioid use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Postoperative chronic pain scores (VAS) at rest and during mobilization | Up to 6 months
  Chronic pain follow-up

SECONDARY OUTCOMES:
Postoperative vital signs | 0-48 hours
  Postoperative early period hemodynamic follow-up
Postoperative acute pain at rest and during coughing/mobilization | 0-48 hours
  Postoperative acute pain score (VAS) follow-up
Postoperative nausea and vomiting (PONV) and antiemetic requirements | 0-48 hours
  Postoperative acute PONV and antiemetic use follow-up
Postoperative morphine consumption | 0-48 hours
  Postoperative IV PCA morphine consumption for Group 1 and IV morphine consumption for Group 2 as rescue analgesic
Time to first analgesic | 0-48 hours
  Postoperative first analgesic IV PCA morphine demand time for Group 1 and first rescue analgesic IV morphine time for Group 2
Postoperative first oral intake, flatulence, defecation, mobilization times | 0-48 hours
  Postoperative first oral intake, flatulence, defecation, mobilization times
Postoperative hospital discharge day and time | Participants is being followed for the duration of hospital stay, an expected average of 1 week
  Postoperative hospital discharge day and time
Postoperative long term (1st, 3rd and 6th months) analgesic, sleep quality and comfort follow-up | Up to 6 months
  Postoperative long term (1st, 3rd and 6th months) analgesic, sleep quality and comfort follow-up with phone call

CONTACTS AND LOCATIONS:
Overall Officials: Mert N Senturk, Prof, Principal Investigator — MD, Prof
Locations (1):
- Istanbul University, Department of Anesthesiology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Komatsu T, Kino A, Inoue M, Sowa T, Takahashi K, Fujinaga T. Paravertebral block for video-assisted thoracoscopic surgery: analgesic effectiveness and role in fast-track surgery. Int J Surg. 2014;12(9):936-9. doi: 10.1016/j.ijsu.2014.07.272. Epub 2014 Aug 1. PMID 25091399